CLINICAL TRIAL: NCT00800722
Title: Phase I Combined Use of Pulsed Dye Laser and Rapamycin
Brief Title: A Randomized Trial to Study Combined Pulsed Dye Laser and Rapamycin Treatment of Port Wine Stain Birthmarks.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Pfizer (Industry); Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, J S Nelson, M.D., Ph.D.,Professor of Surgery and Biomedical Engineering, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20086383.
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Port Wine Stain
Keywords: hypervascular anomalies
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment of Port Wine Stain (Experimental): Rapamycin Treatment of Port Wine Stain
  Interventions: Drug: Rapamycin Treatment of Port Wine Stain

INTERVENTIONS:
Drug: Rapamycin Treatment of Port Wine Stain — Treatment of Port Wine Stain
  Other Names: Treatment of Port Wine Stain

SUMMARY:
The purpose of this study is to improve port wine stain therapeutic outcome in response to laser therapy. The researchers want to determine whether the combined use of pulsed dye laser therapy and rapamycin will improve PWS therapeutic outcome.

DETAILED DESCRIPTION:
The researchers want to combined use of pulsed dye laser to induce port wine stain blood vessel injury, and rapamycin directly inhibits the proliferation of vascular endothelial cells driven by vascular endothelial growth factor which preventing port wine stain angiogenesis and recanalization, to improve port wine stain lesion blanching.

ELIGIBILITY:
Inclusion Criteria:

* port wine stain birthmarks suitable for comparison testing.

Exclusion Criteria:

* Pregnancy.
* Abnormal blood hematology or chemistry blood tests or urine analysis.
* History of cancer, History of high cholesterol, lipids or liver disease
* Allergy to macrolide drugs (e.g., erythromycin).
* Any therapy within the previous two months to the proposed PWS treatment sites.
* Concurrent use of known photosensitizing drugs,immunosuppressive drugs or systemic steroids,antifungals, antiepileptics, HIV protease inhibitors, cimetidine, cisapride, clarithromycin, dannzol, diltiazem, erythromycin, metoclopramide, rifabutin, rifampin, rifapentine, troleandomycin, or verapamil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
improve port wine stain (PWS) therapeutic outcome | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John S Nelson, M.D,PhD, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute Medical clinic, Irvine, California, United States